CLINICAL TRIAL: NCT04824131
Title: Safety, Tolerability and Acceptability of Long-Acting Cabotegravir (CAB LA) for the Prevention of HIV Among Adolescent Females - A Sub-study of HPTN 084
Brief Title: Safety, Tolerability and Acceptability of Long-Acting Cabotegravir (CAB LA) for the Prevention of HIV Among Adolescent Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ViiV Healthcare (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 084-01; 38655 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2021-01-06; First posted 2021-04-01 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAB LA (Experimental): In Step 1, participants will receive one CAB tablet orally every day for 5 weeks. In Step 2, participants will receive an intramuscular (IM) injection of CAB LA at Weeks 5, 9, 17, 25, and 33. In Step 3, participants will receive a TDF/FTC tablet orally every day for 48 weeks or join an open-label extension CAB study in their area, if available.
  Interventions: Drug: Oral cabotegravir (CAB); Drug: CAB LA; Drug: Oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC)

INTERVENTIONS:
Drug: Oral cabotegravir (CAB) — 30 mg tablets
Drug: CAB LA — Administered as one 3 mL (600 mg) IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter
Drug: Oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) — 300 mg/200 mg fixed-dose combination tablets

SUMMARY:
This study will establish the minimum safety, tolerability and acceptability data needed to support the use of cabotegravir long-acting injection (CAB LA) in an adolescent population, potentially transforming the field of HIV prevention for young people.

DETAILED DESCRIPTION:
This study will enroll sexually-active, healthy, HIV-uninfected adolescents assigned female sex at birth. Total participant commitment for the entire study is approximately 1.5 years.

This study will take place in three steps. In Step 1, participants will receive daily oral CAB tablets for 5 weeks. In Step 2, participants will receive a series of five intramuscular (IM) injections of CAB LA, administered at 8-week intervals after a 4-week loading dose (injections at Weeks 5, 9, 17, 25 & 33). A safety visit will follow each injection to ascertain safety data, including injection site reactions. In Step 3, all participants who have received at least one injection will be followed quarterly (every 3 months) for 48 weeks after their last injection. Participants will receive oral TDF/FTC for daily use for 48 weeks or join and open-label extension CAB study in their area, if available.

Participants will attend about 18 study visits throughout the study. Visits may include physical examinations, blood collection, urine collection, vaginal swab collection, risk reduction and adherence counseling, and behavioral or acceptability assessments.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth
* At enrollment, below 18 years of age
* At enrollment, body weight ≥ 35 kg (77 lbs.)
* Willing and able to provide informed assent/consent for the study and/or able to obtain written parental/guardian informed consent
* Self-reported sexual activity with a male (oral, anal or vaginal) in the past 12 months
* Willing and able to undergo all study procedures
* In general, good health, as evidenced by the following laboratory values:

  * Non-reactive / negative HIV test results**,
  * Absolute neutrophil count > 799 cells/mm3,
  * Platelet count ≥ 100,000/mm3,
  * Hemoglobin ≥ 11g/dL,
  * Calculated creatinine clearance ≥ 60 mL/minute using the modified Schwartz equation,
  * Alanine aminotransferase (ALT) < 2.0 times the upper limit of normal (ULN) (≤ grade 1) and total bilirubin (Tbili) ≤ 2.5 x ULN,
  * Hepatitis B virus (HBV) surface antigen (HBsAg) negative) and accepts vaccination,
  * Hepatitis C virus (HCV) Antibody negative
* Must have a negative beta human chorionic gonadotropin (βHCG) pregnancy test (sensitivity of ≤ 25 mIU/mL) performed (and results known) on the same day as Enrollment and before initiating study product
* Must agree to use a reliable form of long acting contraception, during the trial and for 48 weeks after stopping the long acting injectable, or 30 days after stopping oral study product, from the list below:

  * Intrauterine device (IUD) or intrauterine system (IUS) that meets <1% failure rate as stated in the product label
  * Hormone-based contraceptive that meets <1% failure rate when used consistently and correctly as stated in the product label (implants or injectables only; this excludes combined oral contraception)
* If currently on PrEP from a non-study source, willing to stop said PrEP prior to enrollment and agree to switch to oral CAB for the lead-in period and CAB LA injections.
* HIV-uninfected, based on HIV test results obtained at Screening and at the Enrollment visit. All HIV test results from the Screening visit must be obtained and must all be negative/non-reactive. This includes testing for acute HIV infection, which must be performed within 14 days of Enrollment. Individuals who have one or more reactive or positive HIV test result(s) will not be enrolled, even if subsequent confirmatory testing indicates that they are not HIV-infected (see SSP Manual).

Exclusion Criteria:

* Co-enrollment in any other HIV interventional research study or other concurrent studies which may interfere with this study (as provided by self-report or other available documentation)
* Past or current participation in HIV vaccine trial with exception for participants who can provide documentation of receipt of placebo
* Exclusively had sex with biological females in lifetime
* In the last 6 months (at the time of screening):

  * active or planned use of any substance use which would, in the opinion of the site investigator, interfere with study participation (including herbal remedies), as described in the Investigator's Brochure (IB) or listed in the Study Specific Procedures (SSP), and/ or Protocol Section 4.4,
* Known history of clinically significant cardiovascular disease, as defined by history/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease
* Inflammatory skin conditions that compromise the safety of intramuscular (IM) injections
* Tattoo or other dermatological condition overlying the buttock region that may interfere with interpretation of injection site reactions
* Current or chronic history of liver disease (e.g., non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy)
* Known history of clinically significant bleeding
* A history of seizure disorder, per self-report
* Medical, social or other condition that, in the opinion of the site investigator, would interfere with the conduct of the study or safety of the participant (e.g., provided by self-report, or found upon medical history and examination or in available medical records)
* Plans to move out of the geographic area within the next 18 months or otherwise unable to participate in study visits, according to the site investigator
* Pregnant or currently breastfeeding at the time of screening or intends to become pregnant and/or breastfeed while on study

Max Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Study Chair — Stroger Hospital of Cook County; Lynda Stranix-Chibanda, MBChB, MMED, Study Chair — University of Zimbabwe College of Health Sciences
Locations (3):
- Ward 21 CRS, Johannesburg, Gauteng, South Africa
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda
- Spilhaus CRS, Harare, Zimbabwe

REFERENCES:
- [Derived] Stranix-Chibanda L, Hamilton EL, Ngo J, Jiao Y, Hanscom B, Choudhury RP, Agyei Y, Piwowar-Manning E, Marzinke M, Delany-Moretlwe S, Mgodi N, Siziba B, Naidoo I, Gati Mirembe B, Kamira B, McCoig C, Adeyeye A, Spiegel HML, Hosek S; HPTN 084-01 Protocol Team. Safety, tolerability, and acceptability of long-acting injectable cabotegravir for HIV prevention in cisgender female adolescents (HPTN 084-01): a single-arm, open-label, phase 2b trial. Lancet HIV. 2025 Apr;12(4):e252-e260. doi: 10.1016/S2352-3018(24)00310-2. Epub 2025 Mar 12. PMID 40088909

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study target population is sexually-active, healthy female adolescents aged below 18 years. The study target is to enroll more than 50 participants with at least 50 participants receiving at least one injection. Participant recruitment will take approximately 12 months.
Pre-assignment Details: A total of 55 participants were eligible and enrolled. The Study has 3 steps, Oral CAB, Injection CAB LA and the Follow-up of Injection CAB levels with use of TDF/FTC, Truvada® for daily use for 48 weeks. Two participants terminated before Step 2 "Refused participation" and "Adverse Event" so 53 participants received CAB LA injection. Finally out of 53 in Step 3 two further terminated due to " Refused Participation".
Groups:
- Cabotegravir Long Acting: Oral cabotegravir (30mg tablet) Injectable cabotegravir 3 mL (600 mg) intramuscular (IM) injection Oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC): 300 mg/200 mg fixed-dose combination tablets
Period: CAB LA Oral Phase
Arm/Group | Cabotegravir Long Acting
Started (5-week oral CAB 30mg QD) | 55
Completed | 53
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: CAB LA Injection Phase
Arm/Group | Cabotegravir Long Acting
Started (5 intramuscular (IM) injections of 3 mL (600 mg) cabotegravir administered at 8-week intervals after a 4-week loading dose (injections at weeks 5, 9, 17, 25 & 33)) | 53
Completed | 53
Not Completed | 0
Period: Step 3
Arm/Group | Cabotegravir Long Acting
Started (A blood draw visit, the +8 Week Visit, will follow the last injection to monitor CAB drug levels, with additional blood collection at the +24, +36, and +48 Week Visits. Waning levels of cabotegravir (the PK tail) will be covered with locally sourced oral Tenofovir/emtricitabine (Trade name: TDF/FTC, Truvada®) for daily use for 48 weeks) | 53
CAB Open-Label Extension (At "Step 3" participants could either receive oral Tenofovir/emtricitabine OR enter an open-label extension study for Cabotegravir.) | 49 (Two participant completed Step 3 but did not transition to CAB Open-Label Extension)
Tenofovir/Emtricitabine" (At "Step 3" participants could either receive oral Tenofovir/emtricitabine OR enter an open-label extension study for Cabotegravir.) | 0
Completed | 51
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Includes all enrolled participants
Groups:
- Cabotegravir Long Acting: In Step 1, participants will receive one CAB tablet orally every day for 5 weeks. In Step 2, participants will receive an intramuscular (IM) injection of CAB LA at Weeks 5, 9, 17, 25, and 33. In Step 3, participants will receive a TDF/FTC tablet orally every day for 48 weeks or join an open-label extension CAB study in their area, if available.
  Oral cabotegravir (CAB): 30 mg tablets
  CAB LA: Administered as one 3 mL (600 mg) IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter
  Oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC): 300 mg/200 mg fixed-dose combination tablets
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.0 (1.1)
Age, Customized [Count of Participants; unit: Participants]
  12-15 years old | 15
  16-17 years old | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 35
  Shona | 20
Region of Enrollment [Number; unit: participants]
  Uganda | 17
  South Africa | 18
  Zimbabwe | 20
Sexual Orientation: Straight/Heterosexual [Count of Participants; unit: Participants] | 55
Weight [Count of Participants; unit: Participants]
  <50 kg | 15
  >=50 kg | 40
Number of Participants per BMI Category as Determined by Age-Standardized Z-score [Count of Participants; unit: Participants] — Based on age in months. Final z-scores calculated using World Health Organization (WHO) tool https://www.who.int/tools/growth-reference-data-for-5to19-years/indicators/bmi-for-age. Categories allocated according to the following z-scores:
  Obesity: > +2; Overweight: > +1 and <= +2; Normal: > -2 and <= +1; Thinness: > -3 and <= -2; Severe thinness: <= -3.
  Participants
    Obese | 2
    Overweight | 14
    Normal | 38
    Thinness | 1
    Severe thinness | 0

OUTCOME MEASURES:

1. Primary Outcome: Count and Percentage of Participants Experiencing Any Grade 2 or Higher Clinical Adverse Events (AEs) and Laboratory Abnormalities Among Participants Who Receive at Least One Injection of CAB LA.
Description: Number and percent of participants experiencing any Grade 2 or higher clinical adverse events (AEs) or laboratory abnormalities (reported as adverse events) from the first injection visit to 8 weeks after the last Step 2 injection visit or week 41, whichever comes first.
Time Frame: Measured through participant's first injection visit up to, 8 weeks after the last Step 2 injection visit or week 41
Population: Includes enrolled female adolescent participants who receive at least one injection of CAB LA.
Measure: Count of Participants; unit: Participants
Groups:
- Cabotegravir Long Acting: Injectable cabotegravir 3 mL (600 mg) intramuscular (IM) injection
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 53
Participants | 50

2. Primary Outcome: Tolerability Endpoint: Percentage of Participants Who Receive at Least 1 Injection and Who Discontinue Receiving Injections Prior to the Full Course of Injections Due to Intolerability of Injection, Frequency of Injections or Burden of Study Procedures.
Description: Number and percent of participants who receive at least 1 injection and who discontinue receiving injections prior to the full course of injections due to intolerability of injection or burden of study procedures. Reasons for intolerability may include:
  1. Injection site reaction
  2. Burden of study procedure i. Participant refused further participation ii. Participant is unwilling or unable to comply with required study procedures iii. Participant refused further study product use iv. Participant unable to adhere to visit schedule
Time Frame: Measured through participant's first injection visit up to, 8 weeks after the last Step 2 injection visit or week 41
Population: Includes enrolled female adolescents who receive at least one injection of CAB LA.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 53
Participants
  Number of participants who have reported any injection site reaction (ISR) | 14
  Number of participants who have reported any grade 2 (moderate) and above ISR | 3
  Participants who Discontinued Early due to Intolerability of Injection or Burden of Study Procedures | 0
  Enrolled Participants who Completed all Scheduled Injections | 53
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 0.0, 95% CI 2-sided [0 to 6.7]; Exact 95% Confidence Interval for Proportion for Participants who Discontinued Early due to Intolerability of Injection or Burden of Study Procedures

3. Primary Outcome: Acceptability Endpoint: Count and Percentage of Participants Who Complete All Scheduled Injections and Who Receive at Least One Injection Whom Would Consider Using CAB LA for HIV Prevention in the Future.
Description: Number and percent of participants who complete all scheduled injections: Defined as completing all scheduled injections for participants who are confirmed pregnant, confirmed HIV seroconverted, or discontinue product due to the following reasons:
  * Death
  * Early study closure
  * HBV infection
  During Step 1:
  Enrolled population: completed all 0 of 0 scheduled injections Injection population: not applicable, did not receive injection
  During Step 2:
  Both enrolled and injection: completed all injections whose target window closed prior to pregnancy/seroconversion/product discontinuation date
Time Frame: Measured through participant's first injection visit up to, 8 weeks after the last Step 2 injection visit or week 41
Population: Includes enrolled female adolescents who receive at least one injection of CAB LA and who Completed All Scheduled Injections
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 52
Participants
  Participants with Acceptability Endpoint at the end of Step 2 | 52
  Participants who received at least one injection and preferred injectable PrEP at end of Step 2 | 32
  If you wanted to protect yourself from getting HIV: Prefer not using a product | 1
  If you wanted to protect yourself from getting HIV: Condoms only | 7
  If you wanted to protect yourself from getting HIV: Oral PrEP pills only | 1
  If you wanted to protect yourself from getting HIV: Injectable PrEP only | 12
  If you wanted to protect yourself from getting HIV: Condoms and oral PrEP pills together | 8
  If you wanted to protect yourself from getting HIV: Condoms and injectable PrEP together | 20
  If you wanted to protect yourself from getting HIV: Prefer not to answer | 3
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 61.5, 95% CI 2-sided [47.0 to 74.7]; Exact 95% confidence interval for proportion for Participants who received at least one injection and preferred injectable PrEP at end of step 2

4. Secondary Outcome: Count of Participants Above the Protein-adjusted Inhibitor Concentration (90%; PA-IC90) at Each Injection Visit
Description: CAB drug concentrations will be measured in plasma to generate CAB-LA concentration-time profiles among study participants. Measurements will occur at study visits during the injection phase of the study as well as during the pharmacologic "tail" phase. Count of participants for injection visits in which a participant remains above the 1x (0.166 mcg/mL), 4x (0.664 mcg/mL) and 8x (1.33 mcg/mL) PA-IC90. Concentrations above the 3 PA-IC90 are associated with rectal protection in a non-human primate study, and concentrations above the 8x PA-IC90 are expected to be associated with protection in humans.
Time Frame: Measured through participant's first Oral visit up to, 10 weeks after the last Step 2 injection visit or week 41
Population: Includes enrolled female adolescents who receive at least one injection of CAB LA.
Measure: Count of Participants; unit: Participants
Groups:
- Cabotegravir Long Acting: Oral cabotegravir (30mg tablet) Injectable cabotegravir 3 mL (600 mg) intramuscular (IM) injection
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 53
Participants
  <4x PA-IC90 | 0
  4x PA-IC90 - <8x PA-IC90: Injection 1 | 19
  4x PA-IC90 - <8x PA-IC90: Injection 2 | 3
  >8x PA-IC90: Injection 1 | 34
  >8x PA-IC90: Injection 2 | 50
  >8x PA-IC90: Injection 3 | 53
  >8x PA-IC90: Injection 4 | 52
  >8x PA-IC90: Injection 5 | 48

5. Secondary Outcome: Measurement of Pharmacokinetic Parameters, Mean and Associated Deviations of Drug Concentrations at Each Injection Visit.
Description: CAB drug concentrations will be measured throughout the study, and the study team will characterize variability in concentrations at each visit by determining mean concentrations, as well as associated deviations.
Time Frame: Measured through weeks 5, 6, 9, 10, 17, 18, 25, 26, 33, 34, 41 (33 +8)
Population: All study participants who have received at least one injection of CAB-LA
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 53
mcg/mL
  <50 Kg: Week 5: number analyzed (Participants) | 15
  <50 Kg: Week 5 | 7.4 (7.2)
  >=50 Kg: Week 5: number analyzed (Participants) | 38
  >=50 Kg: Week 5 | 5.8 (4.5)
  <50 Kg: Week 6: number analyzed (Participants) | 15
  <50 Kg: Week 6 | 4.4 (2.7)
  >=50 Kg: Week 6: number analyzed (Participants) | 38
  >=50 Kg: Week 6 | 1.7 (1.0)
  <50 Kg: Week 9: number analyzed (Participants) | 15
  <50 Kg: Week 9 | 3.3 (1.7)
  >=50 Kg: Week 9: number analyzed (Participants) | 38
  >=50 Kg: Week 9 | 2.1 (1.6)
  <50 Kg: Week 10: number analyzed (Participants) | 15
  <50 Kg: Week 10 | 5.1 (2.1)
  >=50 Kg: Week 10: number analyzed (Participants) | 38
  >=50 Kg: Week 10 | 3.1 (1.5)
  <50 Kg: Week 17: number analyzed (Participants) | 15
  <50 Kg: Week 17 | 3.2 (0.9)
  >=50 Kg: Week 17: number analyzed (Participants) | 38
  >=50 Kg: Week 17 | 2.9 (1.2)
  <50 Kg: Week 18: number analyzed (Participants) | 15
  <50 Kg: Week 18 | 4.5 (1.3)
  >=50 Kg: Week 18: number analyzed (Participants) | 38
  >=50 Kg: Week 18 | 3.9 (1.6)
  <50 Kg: Week 25: number analyzed (Participants) | 15
  <50 Kg: Week 25 | 3.5 (1.1)
  >=50 Kg: Week 25: number analyzed (Participants) | 38
  >=50 Kg: Week 25 | 3.1 (1.1)
  <50 Kg: Week 26: number analyzed (Participants) | 14
  <50 Kg: Week 26 | 5.0 (1.9)
  >=50 Kg: Week 26: number analyzed (Participants) | 38
  >=50 Kg: Week 26 | 3.8 (1.2)
  <50 Kg: Week 33: number analyzed (Participants) | 14
  <50 Kg: Week 33 | 3.8 (1.3)
  >=50 Kg: Week 33: number analyzed (Participants) | 38
  >=50 Kg: Week 33 | 3.3 (1.1)
  <50 Kg: Week 34: number analyzed (Participants) | 14
  <50 Kg: Week 34 | 4.5 (1.4)
  >=50 Kg: Week 34: number analyzed (Participants) | 38
  >=50 Kg: Week 34 | 4.2 (1.4)
  <50 Kg: Week 42: number analyzed (Participants) | 12
  <50 Kg: Week 42 | 3.7 (1.0)
  >=50 Kg: Week 42: number analyzed (Participants) | 34
  >=50 Kg: Week 42 | 3.2 (1.0)

6. Secondary Outcome: Count and Percentage of Participants Experiencing Grade 2 or Higher Clinical AEs and Laboratory Abnormalities in the Oral Phase and the Aggregate Oral and Injection Phases
Description: Number and percent of participants experiencing any Grade 2 or higher clinical adverse events (AEs) or laboratory abnormalities from:
  1. enrollment to week 5 (oral phase (step 1), including interim visits).
  2. enrollment to 8 weeks following the last injection received (aggregate over oral + injection phases (step 1-step 2) including interim visits)
Time Frame: Measured through participant's first Oral visit up to, 8 weeks after the last Step 2 injection visit or week 41
Population: Includes enrolled female adolescents.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 55
Participants
  Number of Participants with Grade 2 or Higher AEs in Oral Phase | 31
  Number of Participants with Grade 2 or above AEs during Injection Phase: number analyzed (Participants) | 53
  Number of Participants with Grade 2 or above AEs during Injection Phase | 50
  Number of Participants with Grade 2 or Higher AEs in Oral and Injection Phase | 51
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 94.3, 95% CI 2-sided [84.3 to 98.8]; The Exact 95% Confidence Interval for Proportion for Number of Participants with Grade 2 or above AEs during Injection Phase

7. Secondary Outcome: Number and Percent of Injection Visits That Occurred "On-time"
Description: Number and percent of injection visits (up to 5 per participant) that occur "on-time", using the number of injections given as the denominator. This will be presented along with the total number and percent of injections given, among all intended injections (i.e. 5 injections per participant).
Time Frame: Measured through participant's last study visit, up to approximately 1.5 years after study entry.
Population: Participants with at least one Injection
Measure: Number; unit: Number of Injections
Units Other Than Participants: Number of Injections Expected
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 53
Number analyzed (Number of Injections Expected) | 263
Number of Injections
  Number of Injections Given | 263
  Number of Injections given On-time | 228
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; Exact CI for Proportions = 100, 95% CI 2-sided [93.3 to 100]; Exact 95% Confidence Interval for Proportion for Participants who received at least one Injection who Completed All Scheduled Injections

8. Secondary Outcome: Change From Enrollment of Self-reported Sexual Behavior (Number of Sexual Partners) During the Study Period
Description: We will use generalized estimating equations (GEE) with robust variance to model change in self-reported sexual behavior from enrollment (W0) to follow up visits (W4, W5, W9, W17, W25, W33, W+12, W+24, W+36, W+48), with an indicator variable for all on-study visits (i.e. enrollment visit = 0) to measure change in the outcome behavior. We will model count outcomes (number of sexual partners) using a poisson model.
Time Frame: Measured through participant's study visit, up to Week 48 from enrollment.
Population: Includes enrolled female adolescents.
Measure: Mean (Standard Deviation); unit: Number of Sexual Partners
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 55
Number of Sexual Partners
  Enrollment: number analyzed (Participants) | 53
  Enrollment | 3 (6.0)
  Week 4: number analyzed (Participants) | 49
  Week 4 | 2 (5.2)
  Week 4: Change from previous visit: number analyzed (Participants) | 47
  Week 4: Change from previous visit | -1 (5.5)
  Week 4: Change from baseline: number analyzed (Participants) | 47
  Week 4: Change from baseline | -1 (5.5)
  Week 5: number analyzed (Participants) | 45
  Week 5 | 2 (3.1)
  Week 5: Change from previous visit: number analyzed (Participants) | 43
  Week 5: Change from previous visit | 0 (4.0)
  Week 5: Change from baseline: number analyzed (Participants) | 43
  Week 5: Change from baseline | -1 (4.8)
  Week 9: number analyzed (Participants) | 51
  Week 9 | 2 (4.8)
  Week 9: Change from previous visit: number analyzed (Participants) | 44
  Week 9: Change from previous visit | 0 (2.4)
  Week 9: Change from baseline: number analyzed (Participants) | 49
  Week 9: Change from baseline | -1 (4.1)
  Week 17: number analyzed (Participants) | 50
  Week 17 | 2 (5.0)
  Week 17: Change from previous visit: number analyzed (Participants) | 49
  Week 17: Change from previous visit | 0 (1.1)
  Week 17: Change from baseline: number analyzed (Participants) | 48
  Week 17: Change from baseline | -1 (4.3)
  Week 25: number analyzed (Participants) | 52
  Week 25 | 3.1 (6.3)
  Week 25: Change from previous visit: number analyzed (Participants) | 50
  Week 25: Change from previous visit | 1 (5.1)
  Week 25: Change from baseline: number analyzed (Participants) | 50
  Week 25: Change from baseline | 0 (3.1)
  Week 33: number analyzed (Participants) | 49
  Week 33 | 2 (4.4)
  Week 33: Change from previous visit: number analyzed (Participants) | 49
  Week 33: Change from previous visit | -1 (3.9)
  Week 33: Change from baseline: number analyzed (Participants) | 47
  Week 33: Change from baseline | -1 (4.2)
  Step 3 - week + 12: number analyzed (Participants) | 29
  Step 3 - week + 12 | 3 (5.8)
  Step 3 - week + 12: Change from previous visit: number analyzed (Participants) | 29
  Step 3 - week + 12: Change from previous visit | 0 (7.7)
  Step 3 - week + 12: Change from baseline: number analyzed (Participants) | 28
  Step 3 - week + 12: Change from baseline | -1 (8.9)
  Step 3 - week + 24: number analyzed (Participants) | 17
  Step 3 - week + 24 | 6 (13.1)
  Step 3 - week + 24: Change from previous visit: number analyzed (Participants) | 17
  Step 3 - week + 24: Change from previous visit | 3 (12.1)
  Step 3 - week + 24: Change from baseline: number analyzed (Participants) | 17
  Step 3 - week + 24: Change from baseline | 2 (7.4)
  Step 3 - week + 36: number analyzed (Participants) | 12
  Step 3 - week + 36 | 6 (14.3)
  Step 3 - week + 36: Change from previous visit: number analyzed (Participants) | 10
  Step 3 - week + 36: Change from previous visit | -1 (2.6)
  Step 3 - week + 36: Change from baseline: number analyzed (Participants) | 11
  Step 3 - week + 36: Change from baseline | 2 (7.8)
  Step 3 - week + 48: number analyzed (Participants) | 2
  Step 3 - week + 48 | 1 (0)
  Step 3 - week + 48: Change from previous visit: number analyzed (Participants) | 2
  Step 3 - week + 48: Change from previous visit | 1 (0.7)
  Step 3 - week + 48: Change from baseline: number analyzed (Participants) | 2
  Step 3 - week + 48: Change from baseline | 1 (0.7)
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Generalized estimating equations (GEE) with robust variance to model change in self-reported sexual behavior from enrollment (W0) to follow up visits (W4, W5, W9, W17, W25, W33, W+12, W+24, W+36, W+48), with an indicator variable for all on-study visits (i.e. enrollment visit = 0) to measure change in the outcome behavior. We will model count outcomes (number of sexual partners) using a poisson model; Test type: Other; p = 0.1093, poisson model — GEE for Change in Sexual Behavior - Number of Sexual Partners - Visit as Continuous Variable. Difference from baselines in the number of sex partners (vaginal or anal sex) reported in the past month; Mean Difference (Final Values) = -0.2728, 95% CI 2-sided [-0.61 to 0.06], Standard Error of Mean 0.1704 — GEE for Change in Sexual Behavior - Number of Sexual Partners - Visit as Continuous Variable. Difference from baselines in the number of sex partners (vaginal or anal sex) reported in the past month

9. Secondary Outcome: Change From Enrollment of Self-reported Sexual Behavior (Increased Episodes of Vaginal or Anal Sex Without a Condom) During the Study Period
Description: We will use generalized estimating equations (GEE) with robust variance to model change in self-reported sexual behavior from enrollment (W0) to follow up visits (W4, W5, W9, W17, W25, W33, W+12, W+24, W+36, W+48), with an indicator variable for all on-study visits (i.e. enrollment visit = 0) to measure change in the outcome behavior. We will model count outcomes (number of episodes of vaginal sex without a condom) using a poisson model and binary outcomes (any episodes of anal sex without a condom) using a logistic model.
Time Frame: Measured through participant's last study visit, up to approximately 1.5 years after study entry.
Population: Includes enrolled female adolescents.
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 55
Number of Episodes
  Vaginal Sex without a Condom: Enrollment: number analyzed (Participants) | 51
  Vaginal Sex without a Condom: Enrollment | 1 (2.1)
  Vaginal Sex without a Condom: Week 4: number analyzed (Participants) | 47
  Vaginal Sex without a Condom: Week 4 | 2 (11.5)
  Vaginal Sex without a Condom: Week 4: Change from previous visit: number analyzed (Participants) | 45
  Vaginal Sex without a Condom: Week 4: Change from previous visit | 1 (11.3)
  Vaginal Sex without a Condom: Week 4: Change from baseline: number analyzed (Participants) | 45
  Vaginal Sex without a Condom: Week 4: Change from baseline | 1 (11.3)
  Vaginal Sex without a Condom: Week 5: number analyzed (Participants) | 46
  Vaginal Sex without a Condom: Week 5 | 2 (9.8)
  Vaginal Sex without a Condom: Week 5: Change from previous visit: number analyzed (Participants) | 42
  Vaginal Sex without a Condom: Week 5: Change from previous visit | 0 (2.0)
  Vaginal Sex without a Condom: Week 5: Change from baseline: number analyzed (Participants) | 44
  Vaginal Sex without a Condom: Week 5: Change from baseline | 1 (9.7)
  Vaginal Sex without a Condom: Week 9: number analyzed (Participants) | 49
  Vaginal Sex without a Condom: Week 9 | 0 (0.5)
  Vaginal Sex without a Condom: Week 9: Change from previous visit: number analyzed (Participants) | 45
  Vaginal Sex without a Condom: Week 9: Change from previous visit | -2 (9.9)
  Vaginal Sex without a Condom: Week 9: Change from baseline: number analyzed (Participants) | 45
  Vaginal Sex without a Condom: Week 9: Change from baseline | -1 (2.2)
  Vaginal Sex without a Condom: Week 17: number analyzed (Participants) | 48
  Vaginal Sex without a Condom: Week 17 | 1 (1.9)
  Vaginal Sex without a Condom: Week 17: Change from previous visit: number analyzed (Participants) | 47
  Vaginal Sex without a Condom: Week 17: Change from previous visit | 1 (1.9)
  Vaginal Sex without a Condom: Week 17: Change from baseline: number analyzed (Participants) | 45
  Vaginal Sex without a Condom: Week 17: Change from baseline | -1 (1.6)
  Vaginal Sex without a Condom: Week 25: number analyzed (Participants) | 49
  Vaginal Sex without a Condom: Week 25 | 2 (12.8)
  Vaginal Sex without a Condom: Week 25: Change from previous visit: number analyzed (Participants) | 47
  Vaginal Sex without a Condom: Week 25: Change from previous visit | 2 (13.3)
  Vaginal Sex without a Condom: Week 25: Change from baseline: number analyzed (Participants) | 46
  Vaginal Sex without a Condom: Week 25: Change from baseline | 1 (12.8)
  Vaginal Sex without a Condom: Week 33: number analyzed (Participants) | 48
  Vaginal Sex without a Condom: Week 33 | 1 (1.3)
  Vaginal Sex without a Condom: Week 33: Change from previous visit: number analyzed (Participants) | 45
  Vaginal Sex without a Condom: Week 33: Change from previous visit | -2 (13.5)
  Vaginal Sex without a Condom: Week 33: Change from baseline: number analyzed (Participants) | 44
  Vaginal Sex without a Condom: Week 33: Change from baseline | -1 (2.3)
  Vaginal Sex without a Condom: Step 3 - week + 12: number analyzed (Participants) | 29
  Vaginal Sex without a Condom: Step 3 - week + 12 | 1 (2.2)
  Vaginal Sex without a Condom: Step 3 - week + 12: Change from previous visit: number analyzed (Participants) | 27
  Vaginal Sex without a Condom: Step 3 - week + 12: Change from previous visit | 0 (2.2)
  Vaginal Sex without a Condom: Step 3 - week + 12: Change from baseline: number analyzed (Participants) | 27
  Vaginal Sex without a Condom: Step 3 - week + 12: Change from baseline | 0 (3.4)
  Vaginal Sex without a Condom: Step 3 - week + 24: number analyzed (Participants) | 16
  Vaginal Sex without a Condom: Step 3 - week + 24 | 0 (0.7)
  Vaginal Sex without a Condom: Step 3 - week + 24: Change from previous visit: number analyzed (Participants) | 16
  Vaginal Sex without a Condom: Step 3 - week + 24: Change from previous visit | -1 (2.8)
  Vaginal Sex without a Condom: Step 3 - week + 24: Change from baseline: number analyzed (Participants) | 14
  Vaginal Sex without a Condom: Step 3 - week + 24: Change from baseline | -1 (1.9)
  Vaginal Sex without a Condom: Step 3 - week + 36: number analyzed (Participants) | 12
  Vaginal Sex without a Condom: Step 3 - week + 36 | 2 (4.4)
  Vaginal Sex without a Condom: Step 3 - week + 36: Change from previous visit: number analyzed (Participants) | 10
  Vaginal Sex without a Condom: Step 3 - week + 36: Change from previous visit | 2 (4.9)
  Vaginal Sex without a Condom: Step 3 - week + 36: Change from baseline: number analyzed (Participants) | 11
  Vaginal Sex without a Condom: Step 3 - week + 36: Change from baseline | 1 (3.8)
  Vaginal Sex without a Condom: Step 3 - week + 48: number analyzed (Participants) | 2
  Vaginal Sex without a Condom: Step 3 - week + 48 | 0 (0.0)
  Vaginal Sex without a Condom: Step 3 - week + 48: Change from previous visit: number analyzed (Participants) | 2
  Vaginal Sex without a Condom: Step 3 - week + 48: Change from previous visit | -1 (0.7)
  Vaginal Sex without a Condom: Step 3 - week + 48: Change from baseline: number analyzed (Participants) | 2
  Vaginal Sex without a Condom: Step 3 - week + 48: Change from baseline | 0 (0.0)
  Anal Sex without a Condom: Enrollment: number analyzed (Participants) | 50
  Anal Sex without a Condom: Enrollment | 0 (0.0)
  Anal Sex without a Condom: Week 4: number analyzed (Participants) | 46
  Anal Sex without a Condom: Week 4 | 0 (0.2)
  Anal Sex without a Condom: Week 4: Change from previous visit: number analyzed (Participants) | 45
  Anal Sex without a Condom: Week 4: Change from previous visit | 0 (0.2)
  Anal Sex without a Condom: Week 4: Change from baseline: number analyzed (Participants) | 45
  Anal Sex without a Condom: Week 4: Change from baseline | 0 (0.2)
  Anal Sex without a Condom: Week 5: number analyzed (Participants) | 50
  Anal Sex without a Condom: Week 5 | 0 (0.2)
  Anal Sex without a Condom: Week 5: Change from previous visit: number analyzed (Participants) | 44
  Anal Sex without a Condom: Week 5: Change from previous visit | 0 (0.2)
  Anal Sex without a Condom: Week 5: Change from baseline: number analyzed (Participants) | 47
  Anal Sex without a Condom: Week 5: Change from baseline | 0 (0.1)
  Anal Sex without a Condom: Week 9: number analyzed (Participants) | 48
  Anal Sex without a Condom: Week 9 | 0 (0.1)
  Anal Sex without a Condom: Week 9: Change from previous visit: number analyzed (Participants) | 48
  Anal Sex without a Condom: Week 9: Change from previous visit | 0 (0.0)
  Anal Sex without a Condom: Week 9: Change from baseline: number analyzed (Participants) | 46
  Anal Sex without a Condom: Week 9: Change from baseline | 0 (0.1)
  Anal Sex without a Condom: Week 17: number analyzed (Participants) | 50
  Anal Sex without a Condom: Week 17 | 0 (1.1)
  Anal Sex without a Condom: Week 17: Change from previous visit: number analyzed (Participants) | 48
  Anal Sex without a Condom: Week 17: Change from previous visit | 0 (1.2)
  Anal Sex without a Condom: Week 17: Change from baseline: number analyzed (Participants) | 46
  Anal Sex without a Condom: Week 17: Change from baseline | 0 (1.2)
  Anal Sex without a Condom: Week 25: number analyzed (Participants) | 48
  Anal Sex without a Condom: Week 25 | 0 (0.1)
  Anal Sex without a Condom: Week 25: Change from previous visit: number analyzed (Participants) | 47
  Anal Sex without a Condom: Week 25: Change from previous visit | 0 (1.2)
  Anal Sex without a Condom: Week 25: Change from baseline: number analyzed (Participants) | 46
  Anal Sex without a Condom: Week 25: Change from baseline | 0 (0.1)
  Anal Sex without a Condom: Week 33: number analyzed (Participants) | 47
  Anal Sex without a Condom: Week 33 | 0 (0.1)
  Anal Sex without a Condom: Week 33: Change from previous visit: number analyzed (Participants) | 45
  Anal Sex without a Condom: Week 33: Change from previous visit | 0 (0.0)
  Anal Sex without a Condom: Week 33: Change from baseline: number analyzed (Participants) | 44
  Anal Sex without a Condom: Week 33: Change from baseline | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 12: number analyzed (Participants) | 28
  Anal Sex without a Condom: Step 3 - week + 12 | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 12: Change from previous visit: number analyzed (Participants) | 27
  Anal Sex without a Condom: Step 3 - week + 12: Change from previous visit | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 12: Change from baseline: number analyzed (Participants) | 27
  Anal Sex without a Condom: Step 3 - week + 12: Change from baseline | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 24: number analyzed (Participants) | 16
  Anal Sex without a Condom: Step 3 - week + 24 | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 24: Change from previous visit: number analyzed (Participants) | 16
  Anal Sex without a Condom: Step 3 - week + 24: Change from previous visit | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 24: Change from baseline: number analyzed (Participants) | 15
  Anal Sex without a Condom: Step 3 - week + 24: Change from baseline | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 36: number analyzed (Participants) | 10
  Anal Sex without a Condom: Step 3 - week + 36 | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 36: Change from previous visit: number analyzed (Participants) | 9
  Anal Sex without a Condom: Step 3 - week + 36: Change from previous visit | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 36: Change from baseline: number analyzed (Participants) | 9
  Anal Sex without a Condom: Step 3 - week + 36: Change from baseline | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 48: number analyzed (Participants) | 2
  Anal Sex without a Condom: Step 3 - week + 48 | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 48: Change from previous visit: number analyzed (Participants) | 2
  Anal Sex without a Condom: Step 3 - week + 48: Change from previous visit | 0 (0.0)
  Anal Sex without a Condom: Step 3 - week + 48: Change from baseline: number analyzed (Participants) | 2
  Anal Sex without a Condom: Step 3 - week + 48: Change from baseline | 0 (0.0)
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Generalized estimating equations (GEE) with robust variance to model change in self-reported sexual behavior from enrollment (W0) to follow up visits (W4, W5, W9, W17, W25, W33, W+12, W+24, W+36, W+48), with an indicator variable for all on-study visits (i.e. enrollment visit = 0) to measure change in the outcome behavior. We will model count outcomes (number of episodes of vaginal sex without a condom) using a poisson model; Test type: Other; p = 0.0093, poisson model — GEE for Change in Sexual Behavior - Number of Episodes of Vaginal Sex without a Condom - Visit as Continuous Variable. Difference from baselines in the number of vaginal sex without a condom reported in the past month; Mean Difference (Final Values) = -0.5859, 95% CI 2-sided [-1.03 to -0.14], Standard Error of Mean 0.2253 — GEE for Change in Sexual Behavior - Number of Episodes of Vaginal Sex without a Condom - Visit as Continuous Variable. Difference from baselines in the number of vaginal sex without a condom reported in the past month
Statistical Analysis 2: Comparison: Cabotegravir Long Acting; Generalized estimating equations (GEE) with robust variance to model change in self-reported sexual behavior from enrollment (W0) to follow up visits (W4, W5, W9, W17, W25, W33, W+12, W+24, W+36, W+48), with an indicator variable for all on-study visits (i.e. enrollment visit = 0) to measure change in the outcome behavior. We will model binary outcomes (any episodes of anal sex without a condom) using a logistic model; Test type: Other; p = 0.8259, Regression, Logistic — GEE for Change in Sexual Behavior - Number of Episodes of Anal Sex without a Condom - Visit as Continuous Variable. Difference from baselines in the number of anal sex without a condom reported in the past month; Mean Difference (Final Values) = -0.3087, 95% CI 2-sided [-3.06 to 2.44], Standard Error of Mean 1.4036 — GEE for Change in Sexual Behavior - Number of Episodes of Anal Sex without a Condom - Visit as Continuous Variable. Difference from baselines in the number of anal sex without a condom reported in the past month

10. Secondary Outcome: Evaluate Rates of HIV Drug Resistance Among Participants Who Acquire HIV Infection During the Study
Description: Data from steps 1, 2, and 3 will be included. The number of cases of drug resistance will be summarized. All cases of drug resistance among incident HIV infections will be described.
Time Frame: Measured through participant's last study visit, up to approximately 1.5 years after study entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting
Number analyzed (Participants) | 55
Participants
  Total Participants HIV-positive at Enrollment | 0
  Number of participants infected | 0
  Number of drug resistance cases | 0
Statistical Analysis 1: Comparison: Cabotegravir Long Acting; Test type: Other; CI for Incidence rate, exact Poisson = 0.0, 95% CI 2-sided [0.0 to 10.8] — Person-years: 34.0; Incidence rate is calculated HIV infections per 100 person years. CI for Incidence rate is calculated using exact Poisson method

ADVERSE EVENTS:
Time Frame: Measured through participant's first Oral visit up to, follow-up 48 weeks Step 3
Description: SAE, NON SAE & Mortality are summarized by Steps (Oral, Injection & Follow-up).
Groups:
- Step 1 - CAB LA Oral Phase: A 5-week oral CAB 30mg QD safety lead-in
- Step 2 - CAB LA Injection Phase: A series of 5 intramuscular (IM) injections of 3 mL (600 mg) cabotegravir administered at 8-week intervals after a 4-week loading dose (injections at weeks 5, 9, 17, 25 & 33)
- Step 3 - Follow up: A blood draw visit, the +8 Week Visit, will follow the last injection to monitor CAB drug levels, with additional blood collection at the +24, +36, and +48 Week Visits. All participants who have received at least one injection will be followed for 48 weeks after their last injection. Waning levels of cabotegravir (the PK tail) will be covered with locally sourced oral Tenofovir/emtricitabine (Trade name: TDF/FTC, Truvada®) for daily use for 48 weeks.
Arm/Group | Step 1 - CAB LA Oral Phase | Step 2 - CAB LA Injection Phase | Step 3 - Follow up
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/53 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/55 | 2/53 | 0/48
Other Adverse Events (participants affected / at risk) | 48/55 | 52/53 | 29/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Step 1 - CAB LA Oral Phase (N=55) | Step 2 - CAB LA Injection Phase (N=53) | Step 3 - Follow up (N=48)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Step 1 - CAB LA Oral Phase (N=55) | Step 2 - CAB LA Injection Phase (N=53) | Step 3 - Follow up (N=48)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 0 (0) | 3 (4) | 5 (6)
Genitourinary tract gonococcal infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (3)
Gonococcal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 9 (11) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginitis trichomonal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 6 (9) | 1 (1)
Amylase increased (Investigations) | 14 (14) | 19 (27) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 12 (12) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3) | 7 (11) | 2 (2)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 7 (9) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 9 (13) | 2 (2)
Blood glucose decreased (Investigations) | 4 (4) | 20 (27) | 3 (3)
Blood glucose increased (Investigations) | 4 (4) | 21 (27) | 1 (1)
Blood phosphorus decreased (Investigations) | 4 (4) | 6 (8) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 16 (16) | 40 (73) | 4 (4)
Haemoglobin decreased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 11 (11) | 17 (32) | 3 (3)
Low density lipoprotein increased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (6) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 5 (5) | 1 (1)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 8 (15) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 2 (2) | 9 (13) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 2 (2) | 10 (10) | 2 (2)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT04824131/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT04824131/SAP_001.pdf